CLINICAL TRIAL: NCT05524025
Title: Characterizing the Specificity and Sensitivity of Oral TTMV-HPV DNA Testing: The SPOT-HPV Study
Brief Title: The SPOT-HPV Study
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Eleni Marie Rettig, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 22-377
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: HPV Infection; HPV Positive Oropharyngeal Squamous Cell Carcinoma
Keywords: HPV Infection; HPV-positive throat cancer
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A small amount of oral rinse fluid will be banked for future use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Cohort: Adult Male Without HPV-positive throat cancer: Participants will receive 1x Salivary TTMV-HPV DNA Test. If test is negative there will not be follow up, if test is positive participants will have repeat Salivary TTMV-HPV DNA Test, a blood test and head and neck exam.
  Interventions: Diagnostic Test: Salivary TTMV-HPV DNA Test; Diagnostic Test: Blood TTMV-HPV DNA Test
- Case Cohort: Any Adult With HPV-positive throat cancer: Participants will receive 1x Salivary and Blood TTMV-HPV DNA Test(s).
  Interventions: Diagnostic Test: Salivary TTMV-HPV DNA Test

INTERVENTIONS:
Diagnostic Test: Salivary TTMV-HPV DNA Test — Mouthwash rinse
Diagnostic Test: Blood TTMV-HPV DNA Test — Blood test
  Groups: Control Cohort: Adult Male Without HPV-positive throat cancer

SUMMARY:
The purpose of this research is to evaluate a new test for oral HPV DNA in saliva ('oral rinse test').

DETAILED DESCRIPTION:
This cross-sectional study will characterize the prevalence of salivary TTMV-HPV DNA among participants with and without HPV-positive throat cancer

Oral HPV infection is common among healthy adult men, but most of these infections resolve spontaneously and only a very small percentage of oral HPV infections turn into HPV-positive throat cancer. This study is trying to understand whether this new oral rinse test detects HPV DNA from infection, cancer cells, or both. If this test is ONLY positive in people WITH cancer, it may be useful for diagnosing HPV-positive throat cancer in the future.

Along with the oral rinse test study participants will complete brief surveys and participants with a positive salivary TTMV-HPV DNA tests may have repeat saliva testing, blood tests and head/neck exam.

It is expected that about 360 people will take part in this research study.

An external laboratory called Naveris is supporting this research study by providing testing for HPV DNA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years
* Able to provide informed consent
* Either one of the following:

  * Control cohort: Male individuals WITHOUT head and neck tumors that are, or may be, HPV-positive
  * Case cohort: Any individual WITH incident, untreated HPV-positive oropharynx squamous cell carcinoma

Exclusion Criteria:

* Unable to provide informed consent
* Head and neck tumors of non-oropharynx subsites that are or may be HPV-positive, including oral cavity, sinonasal, laryngeal, hypopharyngeal, or nasopharyngeal squamous cell carcinomas

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Control cohort population is adult male
Study Population: Clinic schedules will be screened by the study team to identify eligible participants.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of salivary TTMV-HPV DNA | 12 months
  Percentage of controls without cancer compared with percentage of cancer patients who have TTMV-HPV DNA detected in their saliva

CONTACTS AND LOCATIONS:
Overall Officials: Eleni M Rettig, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham & Woman's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu